CLINICAL TRIAL: NCT04671472
Title: Efficacy Confirmation Study of NPC-09
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPC-09-1
Record Dates: First submitted 2020-11-30; First posted 2020-12-17 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: GNE Myopathy; Distal Myopathy With Rimmed Vacuoles (DMRV); Hereditary Inclusion Body Myopathy (hIBM); Nonaka Disease
Keywords: GNE myopathy; Distal myopathy with rimmed vacuoles (DMRV); Hereditary inclusion body myopathy (hIBM); Nonaka disease; sialic acid; aceneuramic acid; N-acetylneuraminic acid
MeSH Terms: conditions — Distal myopathy, Nonaka type

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aceneuramic acid tablets (Experimental): Aceneuramic acid tablets 6 g/day, divided 3 times a day for 48 weeks
  Interventions: Drug: NPC-09
- Aceneuramic acid placebo tablets (Placebo Comparator): Matching placebo 3 times a day for 48 weeks
  Interventions: Drug: NPC-09 placebo

INTERVENTIONS:
Drug: NPC-09 — The drug will be administered by the oral route with the same manner
  Other Names: Aceneuramic acid tablets
  Arms: Aceneuramic acid tablets
Drug: NPC-09 placebo — The drug will be administered by the oral route with the same manner
  Other Names: Aceneuramic acid matching placebo
  Arms: Aceneuramic acid placebo tablets

SUMMARY:
GNE myopathy is a distal myopathy that is thought to be caused by a mutation in the GNE gene that encodes an enzyme in the biosynthetic process of aceneuramic acid (typical sialic acid). The investigators will examine the efficacy and safety of aceneuramic acid (SA-ER tablets) 6g daily for 48 weeks in patients with GNE myopathy in a placebo-controlled, double-blind, controlled trial.

DETAILED DESCRIPTION:
GNE myopathy is a distal myopathy that is thought to be caused by a mutation in the GNE gene that encodes an enzyme in the biosynthetic process of aceneuramic acid (typical sialic acid). It is an extremely rare progressive muscle disease, often occurring in the late teens to 30s, usually affecting the distal lower leg, especially the extensor muscles such as the tibialis anterior muscle, first, and weakness in both upper and lower limbs. However, the weakness of the quadriceps femoris is usually gradual. Although there are large individual differences, health management and deterioration of QOL will eventually become a problem, and in severe cases, constant assistance is required in daily life.

A double-blind comparative study conducted in Japan provided results suggesting efficacy, but the efficacy could not be confirmed in a large-scale international clinical trial, so this study is decided to be conducted. Oral administration of aceneuramic acid tablets 500 mg (SA-ER tablets) or placebo tablets of the same appearance, 4 tablets at a time, 3 times a day for 48 weeks will be examined for differences in efficacy. The target was a total of 10 cases, 7 cases in the active drug group, and 3 in the placebo group. The amount of change in upper extremity composite score (the sum of the average of the right and left HHD scores for grip, shoulder abductors, elbow flexors and elbow extensors) was used, and the secondary endpoints were the doctor's comprehensive evaluation and the GNE myopathy functional activity scale.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and before any research-related procedures are conducted
* Have a documented diagnosis of GNEM, HIBM, distal myopathy with rimmed vacuoles (DMRV), or Nonaka disease due to previously demonstrated mutations in the gene encoding the GNE/MNK enzyme (genotyping will not be conducted in this study)
* Male or female, aged 18 - 50 years at Screening
* Those who have a score of 24 points or more on the upper limbs of GNEM-FAS (GNE Myopathy Functional Activity Scale) and a disease period of 5 years or more and 15 years or less
* Those whose upper limb muscle weakness has been confirmed from the results of manual muscle testing or grip strength measurements over the past few years, or if he / she has participated in the previous clinical trial*, those who could confirm the upper extremity composite score decreased during the investigational drug is not administered.
* Able to provide reproducible force in elbow flexors (i.e. two dynamometry force values with no more than 15% variability in the dominant arm) at Screening
* Willing and able to comply with all study procedures
* Participants of child-bearing potential or with partners of child-bearing potential who have not undergone a bilateral sapling-oophorectomy and are sexually active must consent to use an effective method of contraception as determined by the site investigator (i.e. oral hormonal contraceptives, patch hormonal contraceptives, vaginal ring, intrauterine device, physical double-barrier methods, surgical hysterectomy, vasectomy, tubal ligation or true abstinence) from the period following the signing of the informed consent through 3 months after last dose of study drug
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study.
* Females considered not of childbearing potential include those who have been in menopause for at least two years, have had tubal ligation at least one year prior to Screening, or who have had a total hysterectomy or bilateral salpingo-oophorectomy
* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and before any research-related procedures are conducted

Exclusion Criteria:

* Ingestion of N-acetyl-D-mannosamine (ManNAc), SA, or related metabolites; intravenous immunoglobulin (IVIG); or anything that can be metabolized to produce SA in the body within 60 days prior to the Screening Visit
* Has had any hypersensitivity to the investigational drug (SA-ER or its excipients) that, in the judgment of the investigator, places the subject at increased risk for adverse effects
* History of more than 30 days treatment with SA-ER and/or SA-IR in prior clinical trials in the past year
* Has serum transaminase (i.e. aspartate aminotransferase [AST] or gamma-glutamyl transpeptidase [GGT]) levels greater than 3X the upper limit of normal (ULN) for age/gender, or serum creatinine of greater than 2X ULN at Screening
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or anticipated requirement for any investigational agent prior to completion of all scheduled study assessments
* Has a condition of such severity and acuity, in the opinion of the investigator, that it warrants immediate surgical intervention or other treatment or may not allow safe participation in the study
* Has a concurrent disease, active suicidal ideation, or other condition that, in the view of the investigator, places the subject at high risk of poor treatment adherence or of not completing the study, or would interfere with study participation or would affect safety
* More than 400 mL blood donation within 16 weeks
* Presence of alcohol or drug dependency
* Those whom the investigator judges not to be appropriate for the subject

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the upper extremity composite score (the sum of the average of the right and left muscle strength measured by HHD (Hand held dynamometer) (kg) for grip, shoulder abductors, elbow flexors and elbow extensors) | Week 48
  Muscle strength based on the maximum voluntary isometric contraction (MVIC) is measured.

SECONDARY OUTCOMES:
The effective rate in comprehensive judgement by the investigator | Week 48
  The investigator judges based on below 1 ~ 4 items.
  1. The manual muscle testing (0 - 5) or grip strength (kg)
  2. the upper extremity composite score (kg)
  3. the change in the upper extremity composite score (kg) compared with the transition of non-active drug administered GNE myopathy patients
  4. the other secondary endpoints
Change from Baseline in GNE Myopathy Functional Activity Scale (GNEM-FAS) upper extremity domain score | Week 48
  Upper extremity functional activity is assessed using the upper extremity domain sore of the GNEM-FAS instrument. It consists of 8 items (score 0-4 for each item), total domain score is 0 to 32 with higher scores representing greater activity.
Changes from Baseline in Individual muscle strength: Grip, shoulder abductors, elbow flexors, and elbow extensors comprising the upper extremity composite score (kg) | Week 48
  Muscle strength based on the maximum voluntary isometric contraction (MVIC) is measured.
Change from baseline in knee extensors muscle strength (kg) | Week 48
  Muscle strength based on the maximum voluntary isometric contraction (MVIC) is measured.
Change from Baseline in GNE Myopathy Functional Activity Scale (GNEM-FAS) mobility domain score | Week 48
  Mobility functional activity is assessed using the mobility domain sore of the GNEM-FAS instrument. It consists of 10 items (score 0-4 for each item), total domain score is 0 to 40 with higher scores representing greater activity.
Change from Baseline in GNE Myopathy Functional Activity Scale (GNEM-FAS) self-care domain score | Week 48
  Self-care functional activity is assessed using the self-care domain sore of the GNEM-FAS instrument. It consists of 7 items (score 0-4 for each item), total domain score is 0 to 28 with higher scores representing greater activity.

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka University Hospital, Suita, Osaka
  - National Center Hospital of Neurology and Psychiatry Hospita, Kodaira, Tokyo
  - Kumamoto University Hospital, Kumamoto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mori-Yoshimura M, Suzuki N, Katsuno M, Takahashi MP, Yamashita S, Oya Y, Hashizume A, Yamada S, Nakamori M, Izumi R, Kato M, Warita H, Tateyama M, Kuroda H, Asada R, Yamaguchi T, Nishino I, Aoki M. Efficacy confirmation study of aceneuramic acid administration for GNE myopathy in Japan. Orphanet J Rare Dis. 2023 Aug 11;18(1):241. doi: 10.1186/s13023-023-02850-y. PMID 37568154